CLINICAL TRIAL: NCT03825575
Title: Sacral Neuromodulation as Treatment for Fecal Incontinence
Acronym: LLLT-FI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jihong Chen, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McMasterChenFI
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Anorectal manometry
MeSH Terms: conditions — Fecal Incontinence | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incontinence and low level laser therapy (Experimental): Intervention: Low level laser therapy (sacral neuromodulation or photobiomodulation) will be administered to patients with fecal incontinence
  Interventions: Device: Low level laser therapy (LLLT)

INTERVENTIONS:
Device: Low level laser therapy (LLLT) — A 3 week treatment period with a total of 8 treatments of 1 hour over the sacral spinal cord
  Other Names: Sacral neuromodulation; Photobiomodulation; BioFlex laser stimulation

SUMMARY:
The objective of this study is to investigate if low level laser therapy will do more good than harm for patients with severe refractory fecal incontinence. It is a proof of concept study without a placebo arm.

DETAILED DESCRIPTION:
The therapy consists of a 3 week treatment with a total of 8 sessions of low level laser therapy. Effects will be assessed using symptoms and quality of life questionnaires and physiological assessments of pelvic floor function, at 4 weeks and 12 weeks after beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with fecal incontinence

Exclusion Criteria:

* Pregnant patients
* Known malignancies in the area of treatment
* Active bleeding in area of treatment
* Active deep vein thrombosis
* When tatoos are present at area of treatment
* Patients that are light sensitive
* Patients who take steroids.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-08 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of fecal incontinence episodes | 4 weeks and 12 weeks
  Number of fecal incontinence episodes per week

SECONDARY OUTCOMES:
Change in Quality of Life | 4 weeks and 12 weeks
  The Fecal Incontinence Quality of Life Assessment is a subject-completed questionnaire. It is measured in each of four areas of depression/self-perception (7 items), lifestyle (10 items), coping (9 items), and embarrassment (3 items). Area scores are measured on a 1 (worse) to 4 (best) scale and are each the average of their component individual item scores measured on the same scale. The total score is the mean of all non-missing items. A negative change from baseline indicates improvement. Minimum important difference is 4 (Forte et al., 2016)
Change in symptoms score | 4 and 12 weeks
  St. Mark's Incontinence (Vaizey) Score, it is a scale from 0-24 where 0=perfect continence and 24 is complete continence. Minimal important difference is 3 (Forte et al., 2016)
Change in anal sphincter tone | 12 weeks
  Anal sphincter tone (mmHg)
Change in increase of anal sphincter pressure during squeezing | 12 weeks
  Difference between anal sphincter squeeze pressure and resting pressure (mmHg)
Change in squeezing duration | 12 weeks
  Anal sphincter sustained squeezing duration (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Chen, MD PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forte ML, Andrade KE, Butler M, Lowry AC, Bliss DZ, Slavin JL, Kane RL. Treatments for Fecal Incontinence [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2016 Mar. Report No.: 15(16)-EHC037-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK356097/ PMID 27099893
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117